CLINICAL TRIAL: NCT06923228
Title: A Single-Blind, Prospective Clinical Study to Assess the Efficacy, Safety and Tolerability of CGB-500 1% Tofacitinib Ointment vs. an Active Comparator for Atopic Dermatitis
Brief Title: A Study to Assess Efficacy and Safety of CGB-500, 1% Tofacitinib Versus an Active Comparator for Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CGB-500-05
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tofacitinib; ruxolitinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CGB 500 ointment with 1% tofacitinib (Experimental): topical ointment
  Interventions: Drug: CGB-500 Ointment with 1% tofacitinib
- ruxolitinib cream QD (Active Comparator): topical cream
  Interventions: Drug: Ruxolitinib 1.5% Cream QD

INTERVENTIONS:
Drug: CGB-500 Ointment with 1% tofacitinib — experimental drug
  Arms: CGB 500 ointment with 1% tofacitinib
Drug: Ruxolitinib 1.5% Cream QD — topical cream
  Arms: ruxolitinib cream QD

SUMMARY:
The goal of this clinical trial is to learn if drug CGB-500 works to treat atopic dermatitis in subjects 12 years of age or older. It will also learn about the safety of CGB-500. The main questions it aims to answer are:

Does CGB-500 decrease the severity of atopic dermatitis on the skin? What medical problems do participants have when taking drug CGB-500? Researchers will compare CGB-500 to a an approved product (1.5% ruxolitinib) to see if CGB-500 works to treat atopic dermatitis.

Participants will:

Apply CGB-500 and ruxolitinib to different locations on their body twice a day for four weeks.

Visit the clinic six times for checkups and tests Keep a diary of their symptoms and when they apply the product

ELIGIBILITY:
Inclusion Criteria:

Outpatient, male or female of any race, 12 years of age or older. Females of childbearing potential (FOBCP) must have a negative urine pregnancy test at Screening and Baseline and practice a reliable method of contraception throughout the trial.

2. Have a clinical diagnosis of atopic dermatitis (AD) for at least 12 months prior to Baseline that has been clinically stable disease for ≥ 3 months at the time of the screening visit and prior to dose administration and is confirmed to be AD according to the criteria of Hanifin and Rajka 3. Have an Investigator Global Assessment (IGA) score of 3 (moderate) at Screening and Baseline, conducted for both sides of the body.

4. Have AD lesions/symptoms covering at least 2% but less than 20% of total body BSA (excluding scalp, genitalia, palms, and soles) at Screening and Baseline.

5. Have at least 2 distinct "target treatment areas," one on the right side of the body and one on the left, each covering ≥1% but ≤10% BSA at Screening and Baseline. Multiple target areas are acceptable on each side of the body. Target treatment areas must be representative of the participant's disease state and not be located on the scalp, genitalia, palms, or soles.

6. In general, good health as determined by medical history and physical examination at the time of screening (investigator discretion).

7. Have Peak Pruritus Numeric Rating Scale (PPNRS) score of ≥ 4 on the scale 0 to 10 at Screening and Baseline, assessed for both sides of the body.

8. Be able to follow trial instructions and likely to complete all required visits.

9. Sign the Institutional Review Board/Independent Ethics Committee (IRB/IEC)-approved informed consent form (ICF, which includes HIPAA) and assent prior to any trial-related procedures being performed.-

Exclusion Criteria:

1 Females who are pregnant, breastfeeding, intending to be pregnant during the trial, or who do not agree to use an acceptable form of birth control during the trial if of childbearing potential 2. Immunocompromised individuals as adjudicated by the principal investigator (PI) based on review of medical history.

3. Known hypersensitivity or previous allergic reaction to any constituent of the IP (e.g., tofacitinib or Janus kinase [JAK] inhibitors, essential oils, choline, phosphatidylcholine, glycerol, propylene glycol, polyethylene glycol).

4. Clinically significant safety labs (hematology, chemistry, and urinalysis) at the Screening visit that, in the opinion of the investigator, would preclude participation in the study or affect proper assessment of the study endpoints.

5. Skin infections (e.g., bacterial, fungal or viral) or conditions that can interfere with reliable AD assessments.

6. Basal cell carcinoma within 6 months prior to Baseline. 7. History of significant skin conditions, e.g., psoriasis, rosacea, erythroderma, or ichthyosis or presence of Netherton's Syndrome, immunological deficiencies or diseases, HIV, uncontrolled diabetes, malignancy, or serious active or recurrent infection.

8. Participants who have previously failed or had an inadequate response to oral, systemic or topical JAK inhibitors, including in a trial or under a prescription for AD (e.g., ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, pacritinib).

9. Use within 14 days prior to Baseline of: 1) systemic antibiotics, 2) calcipotriene or 3) retinoids.

10. Has known hepatic impairment or disorder with aspartate aminotransferase (AST)/alanine amino transferase (ALT) > 3x upper limit of normal (ULN) at Screening.

11. Has unstable and impaired renal function with an estimated glomerular filtration rate (eGFR) <60 mL/min using Cockcroft-Gault (C-G) equation (eGFR between 60 to <90 mL/min or higher is acceptable; Section 13.2).

12. Use within 4 weeks prior to Baseline of moderate to strong CYP3A4 and CYP3A5 inhibitors (e.g. ritonavir, clarithromycin, itraconazole, erythromycin, fluconazole, verapamil, ketoconazole, nefazodone, nelfinavir, diltiazem, ciprofloxacin, grapefruit juice).

13. Use within 7 days on the treatment area(s) prior to Baseline of: 1) topical antihistamines, 2) topical antibiotics, 3) topical corticosteroids or 4) other topical drug products.

14. Use of the following treatments prior to Baseline:

1. For 5 half-lives or 12 weeks (whichever is longer) - biologic agents (e.g., dupilumab).
2. For 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs, cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (e.g., mycophenolate or tacrolimus).
3. For 2 weeks - UVA/UVB therapy, PUVA (psoralen plus ultraviolet) therapy, tanning booths, or non-prescription UV light sources.
4. For 2 weeks - immunizations and sedating antihistamines unless on long-term stable regimen (nonsedating antihistamines are permitted).
5. For 2 weeks - use of other topical treatments for atopic dermatitis (other than bland emollients). Diluted sodium hypochlorite "bleach" baths are allowed if they do not exceed 2 baths per week and their frequency remains the same throughout the trial.

   15. Uncontrolled systemic disease, including Hepatitis B and Hepatitis C. 16. Any illness or condition(s) (including any skin or cardiovascular condition) that, in the opinion of the PI, would interfere with full participation in the trial, including administration of IP and attending required trial visits; pose a significant risk to the participant; or interfere with interpretation of trial data.

   17. Foreseen unprotected and intense/excessive UV exposure during the trial. 18. Scheduled or planned surgical procedures during the trial. 19. Unable or unwilling to comply with any of the trial requirements. 20. Medical or psychiatric conditions, or a personal situation, that may increase the risk associated with trial participation or may interfere with interpretation of trial results or participant compliance and, in the opinion of the PI, makes the participant inappropriate for trial entry.

   21. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.

   22. Employees of the research center or Investigator. 23. Family of members of employees of the research center or Investigator. 24. Participants (e.g. siblings, spouses, relatives, roommates) residing in the same household cannot be enrolled at the same time.

   25. Previous participation in a CGB-500 clinical study or exposure to CGB-500. Participants who have previously received CGB-500 as part of any clinical trial or investigational study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
evaluate effectiveness | From enrollment to end of study at 4 weeks
  To evaluate percent change in localized eczema area severity by using the Localized Eczema Area Severity Index (L-EASI) score from Baseline to week 4.
Safety and tolerability | From enrollment to end of study at 4 weeks
  Overall Incidence of safety events tabulated using the current version of the medical dictionary for regulatory activities (MedDRA).

IPD SHARING:
Plan to Share IPD: No